CLINICAL TRIAL: NCT05794386
Title: SCAR Burden of Left Atrium Guided cathEter Ablation sTrategy for Persistent Atrial Fibrillation (SCARLET-AF Study)
Brief Title: SCAR Burden of Left Atrium Guided cathEter Ablation sTrategy for Persistent Atrial Fibrillation
Acronym: SCARLET-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCARLET-AF
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a 1:1 randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PVI only group (No Intervention): Patients will receive PVI alone regardless of LVA burden.
- Additional LA substrate modification group (Experimental): Patients will receive PVI plus additional LA substrate modification according to their LVA burden.
  Interventions: Procedure: LVA-guided LA substrate modification

INTERVENTIONS:
Procedure: LVA-guided LA substrate modification — The LVA-guided additional LA ablation is included linear ablation or LVA zone border modification/isolation/ homogenization. The additional ablation strategies are finally selected at the physicians' discretion, considering LVA location and distribution.
  Arms: Additional LA substrate modification group

SUMMARY:
This is a multicenter, randomized controlled trial to compare the recurrence of 1-year atrial arrhythmia after catheter ablation of atrial fibrillation (AF) between pulmonary vein isolation (PVI) and PVI with additional left atrial (LA) substrate modification based on the left atrial low-voltage area (LA LVA) in patients with persistent AF who had a moderate burden of LVA in LA (1cm2 to <30%).

DETAILED DESCRIPTION:
* Sample size calculation To calculate the sample size needed to conduct the study, the investigators used the test for two proportions. The participants will be 1:1 randomized. Group sample sizes of 91 in group 1 and 91 in group 2 achieve 80.318% power to detect a difference between the group proportions of -0.20. The proportion in group 1 (the treatment group) is assumed to be 0.50 under the null hypothesis and 0.30 under the alternative hypothesis. The proportion in group 2 (the control group) is 0.50. The test statistic used is the two-sided Z-Test with unpooled variance. The significance level of the test is 0.05. When the investigators set the expected drop-out rate as 10%, the final sample size of each group is 102.
* Statistical analysis

  1. Part 1. Randomized controlled trial for LVA burden 1cm2 to <30%

     * Primary endpoint The survival analysis of AT/AF recurrence during 1-year follow-up after the procedure with 3-months of blanking period is performed by Kaplan-Meier survival analysis. The log-rank test compares the survival curve of two groups (PVI only vs. PVI with additional LA substrate modification). To evaluate the effect of LA substrate modification on the recurrence of AT/AF, Cox proportional hazard regression analysis with the log-rank test is performed.
     * Secondary endpoint Kaplan-Meier survival analysis is performed for the recurrence of AT/AF within 3 months, the recurrence of AF or AT between 3 months and one year after the procedure, and a log-rank test will be used to compare the survival curves of the two groups. To evaluate the effect of LA additional substrate modification on the early recurrence of AT/AF within 3-month, and the recurrence of AF or AT between 3 months and 1 year after the procedure, a Cox proportional hazard regression analysis with a log-rank test will be performed. The comparison of the EHRA symptom grade change before and after the procedure and the quality of life evaluation score according to the SF-36 questionnaire before and after the procedure will be analyzed using the paired t-test.
  2. Part 2. Registry for LVA burden <1cm2 or ≥30% Part 2 is classified into <1cm2 group and ≥30% group according to LVA burden, and primary/secondary endpoints are collected in each group. The entire groups are

  <!-- -->

  1. LVA burden 1cm2 to <30%, PVI only group
  2. LVA burden 1cm2 to <30%, PVI + additional LA substrate modification group
  3. LVA burden <1cm2 with PVA only group
  4. LVA burden ≥30% with PVI + additional LA substrate modification group The investigators analyzed the difference in the occurrence of the primary and secondary endpoints in the four groups using the Kaplan-Meier survival analysis and log-rank test. In addition, factors related to the recurrence of AT/AF are analyzed through univariable and multivariable Cox proportional hazard analysis.
* Study Procedures

  1. Subject screening Patients with persistent AF are screened for study enrollment during the outpatient clinic. Patients must receive appropriate anticoagulant treatment for at least 1 month prior to AF catheter ablation.
  2. Informed consent After AF ablation, informed consent for the study is acquired.
  3. Voltage mapping and randomization AF ablation is performed using a 3D mapping system (CARTO). Before the ablation, LA voltage mapping was first performed in sinus rhythm. If a patient's rhythm is not in AF, then electrical cardioversion is performed to restore sinus rhythm and perform voltage mapping. To ensure a sufficient quality of the voltage map, at least 2500 points should be acquired with TPI(Tissue Proximity Index) function On.

After the mapping, the LVA burden is calculated. If the LVA burden is between ≥1cm2 and <30%, the patient is randomized either to the control group (Group 1; PVI alone) or the experimental group (Group 2; PVI alone + LVA burden guided substrate modification).

The participants with the LVA burden <1cm2 or ≥30% will be excluded from the randomization but allocated to the registry. They are not primarily involved in data analysis of the RCT, but their data will be monitored for a further study. We recommend PVI alone for those with the LVA burden <1cm2. For the participants with the LVA burden ≥30%, additional ablation beyond PVI is at physician's discretion.

* Ablation protocol The pre-defined ablation protocol for each group is as follows.

  1. Group 1: PVI alone - The control group The participants in Group 1 received the usual PVI alone. A detailed PVI protocol is as follows.

     * Point-by-point AI(ablation index) guided PVI is performed
     * AI target: 400~500 for roof/anterior sides, 300~400 for posterior/ inferior/ carina sides
     * Ablation power: 30~40 W for roof/anterior sides, 25~45 W for posterior/ inferior/ carina sides
     * Contact force: target 10~20 g
     * VisiTag setting: 2.5 mm, 5 s, 3 g
     * Both exit and entrance blocks should be checked for successful PVI
     * Esophageal temperature monitoring: Not mandatory. If performed, ablation should be immediately stopped if the temperature rises ≥38 ℃
     * Definition of successful PVI: The ablation procedure will be considered successful when PVI, as confirmed by the bidirectional conduction block between PV and LA, has been achieved. A bidirectional conduction block is defined as the combination of an entrance block (the stable absence of conduction into the PV from the LA) and exit block (the stable absence of conduction from the PV into the LA, either spontaneous or during pacing from the circular mapping catheter positioned at the PV ostium).
  2. Group 2: PVI + LVA burden guided substrate modification - The experimental group The participants in Group 2 received usual PVI plus additional LVA burden guided substrate modification. A PVI procedure is same as in Group 1. A detailed protocol for LVA burden guided ablation and its endpoints are as follows.
* LVA burden guided substrate modification

  * Only LVA island(s) ≥1 cm2 should be ablated
  * LVA near PV ostium: PVI ablation should be designed to included the LVA
  * LVA at anterior side: Anterior linear ablation including the LVA is performed
  * LVA at posterior side: Posterior wall isolation including the LVA is performed. If LVA island(s) is small such that focal ablation can be also considered, either posterior wall isolation or focal ablation can be performed by the physician's discretion.
  * LVA at septal or lateral side: Focal homogenization of the LVA is performed
* Endpoints for LVA burden-guided substrate modification

  * Focal ablated LVA: Loss of capture by 10 V, 2 ms.
  * Linear ablation-related LVA: Bidirectional block across the line After the ablation according to the pre-defined protocol, an AF induction test and AF trigger search are performed. Additional ablation can be performed according to the results of the tests.
* Follow-up method 14-day ambulatory ECG monitoring (14-day for RCT, 1- or 3-day for Registry participants).

This study uses a single-lead ECG patch device for the detection of the recurrence of atrial tachyarrhythmia during the follow up. The ECG patch device is capable of 14-day ambulatory ECG monitoring. Compared to 24- or 72-hr Holter test, the use of 14-day ECG monitoring allows for a more accurate examination of the efficacy of the treatment. Additionally, the patient can activate the device manually to facilitate the analysis of heart rhythm during symptomatic events. Arrhythmia events meeting these criteria are stored for independent adjudication by an independent, blinded clinical endpoint committee.

* Follow-up and procedure endpoint evaluation After the ablation, participants will be discharged within 24 hours after the ablation procedure. Participants will be instructed to record symptomatic episodes via the use of the patient activator. Scheduled follow-up visits will occur at 3, 6, and 12 months from the first ablation procedure (within a 4-week margin). After the 90-days of the blanking period, any atrial tachyarrhythmias will be followed up at 3, 6, and 12 months after the procedure. The recurrence can be confirmed by 12-lead ECGs (3, 6, and 12 months) and ambulatory 14-day single-lead ECG monitoring (3, 12 months). Arrhythmia recurrence during the first 90 days blanking period can be treated with cardioversion and/or AADs. Where possible, repeat ablation procedures will be deferred until after the 3-month blanking period due to the potential for a delayed cure (as per standard practice and in accordance with HRS/ECAS/EHRA recommendations). If AADs (except amiodarone) are used in the first 3 months post-ablation, they will be discontinued five half-lives before the end of the 3-month blanking period with the discretion of the operator. After a 3-month post-ablation, the redo procedure would be decided on the discretion of the physician.
* Study discontinuation and withdrawal criteria Research participants have the right to refuse participation in research or to withdraw participation at any time for any reason. In case of refusal or withdrawal from participation in the study, there is no harm, and no future medical management is affected. The researcher may suspend or exclude a participant from the study if at least one of the reasons described below exists.

  * In case of withdrawal of the consent by participants or legal representatives
  * In case of adverse effects related to the study make it difficult to continue the study
  * In case of any violations of inclusion or exclusion criteria are found during the study participation
  * If a researcher judges that continuing the study is difficult
* Risks and Benefits Radiofrequency catheter ablation is commonly used for the treatment of AF. However, different risks could be observed by different ablation strategies. According to the ERASE-AF trial, additional LVA-guided ablation resulted in complications as follows. The investigators assume similar complication rates will be observed in our study.

  * Cardiac tamponade or pericardial effusion: 2.7%
  * Sepsis: 0.3%
  * Femoral arteriovenous fistula: 0.9%
  * Femoral pseudoaneurysm: 2.2%
  * There was no reported stroke/TIA/arterial embolism, pericarditis, phrenic nerve palsy, internal bleeding, atrioesophageal fistula, pulmonary vein stenosis, or death.
  * Compared to the ERASE-AF trial, femoral puncture related complications can be prevent in our study by using sono-guided procedure.

ELIGIBILITY:
Ages eligible for the study: 19 years or older

Inclusion criteria:

1. Patients with symptomatic persistent AF who undergo AF catheter ablation due to continued AF even after anti-arrhythmic agents or
2. Patients with a burden of LA LVA (scar zone) of 1cm2 or more and less than 30% in 3D voltage mapping before the index catheter ablation are included in the randomized assignment group when performing catheter ablation in satisfaction with 1)

4) Patients with an LVA of <1cm2 or ≥30% are recruited as a registry.

Exclusion criteria:

1. Patients with LA anteroposterior diameter of more than 55 mm
2. Patients with prior AF-related catheter ablation or surgery
3. Patients whose exact LVA burden cannot be calculated because high-quality 3D voltage mapping cannot be obtained during the procedure.
4. Inability or unwillingness to receive anticoagulation (heparin or oral anticoagulation)
5. Known severe left ventricular systolic dysfunction (ejection fraction <35%)
6. Patients with severe structural heart disease (severe mitral regurgitation, hypertrophy cardiomyopathy, other severe valvular heart diseases)
7. Patients with intracardiac thrombus
8. Patients with prior cardiac surgery
9. Patients who had a myocardial infarction or underwent percutaneous coronary intervention within three months
10. Patients who had a stroke or transient ischemic attack within 6 months
11. Patients who had a planned operation or procedure for the cardiovascular system
12. Patients with intractable hypertension or uncontrolled thyroid disease
13. Patients who need dialysis due to end-stage renal disease or who are scheduled for dialysis
14. Patients who are currently pregnant or are likely to be pregnant within the study period
15. Patients who are taking immunosuppressive drugs or had undergone chemotherapy for cancer, autoimmune disease, transplant, etc
16. Patients whose life expectancy is less than 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Late recurrence of AT/AF | From 3 months to 1 year after the catheter ablation
  Recurrence of atrial tachyarrhythmia (AT/AF) from 3 months to 1 year after the index procedure

SECONDARY OUTCOMES:
Early recurrence of atrial tachyarrhythmia | Within 3 months from the catheter ablation
  Early recurrence of atrial tachyarrhythmia within 3 months after the index procedure
Late recurrence of AF | From 3 months to 1 year after the catheter ablation
  AF recurrence from 3 months to 1 year after the index procedure
Late recurrence of AT | From 3 months to 1 year after the catheter ablation
  Atrial tachycardia (AT) recurrence from 3 months to 1 year after the index procedure
5. AF-related Quality of Life | Before (at baseline) and after (at 1 year) the catheter ablation
  AF-related quality of life was measured by a survey (AFEQT) performed before and after the index procedure. The AFEQT survey measures scores (lower scores for a better quality of life). The decrement in AFEQT survey scores after the index procedure confirms the better quality of life after the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No